CLINICAL TRIAL: NCT01540929
Title: A Phase IV Post-licensure DOD Screening Accuracy Study in Military Personnel
Brief Title: Post-licensure Department of Defense (DOD) Screening Accuracy Study in Military Personnel
Status: Completed | Type: Observational
Sponsor: Emergent BioSolutions (Industry)
Responsible Party: Sponsor
Other Study IDs: H-406-002; U1111-1122-1978 (Other: WHO)
Record Dates: First submitted 2012-02-23; First posted 2012-02-29 (Estimated); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Smallpox
Keywords: Smallpox; ACAM2000®; Smallpox vaccine
MeSH Terms: conditions — Smallpox

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study Group: DoD Smallpox Screening Form 600 (2 part format)

SUMMARY:
This is a retrospective study of the Department of Defense (DoD) Smallpox Screening Form 600s (SF600s) generated during screening of service members for possible immunization with the ACAM2000® smallpox vaccine.

Primary Objective:

* To evaluate the accuracy of the DoD smallpox vaccination screening process in military personnel.

Secondary Objective:

* To describe the number of subjects who are excluded from vaccination, stratified by the pre-defined categories for exclusion (separately for the Screened and Evaluable Populations).

DETAILED DESCRIPTION:
Please note that we elected to post this study on the registry (clinicaltrials.gov) in the interests of transparency and because the study represented a post-licensure commitment to FDA for ACAM2000® smallpox vaccine. However, this study was not a clinical trial and did not involve the administration of any vaccine product nor the collection of any product performance or adverse event data. Rather, the purpose of the study was to determine the success rate for proper completion and use of Department of Defense (DoD) Screening Form 600s (SF600s). The SF600 is a form required to be completed prior to smallpox vaccination of DoD staff and is used to guide decision-making by DoD vaccination staff regarding offering, postponing, or denying vaccination. The study evaluated both the extent to which the SF600s were completed correctly and the extent to which they were correctly used to guide vaccination decision-making.

ELIGIBILITY:
Inclusion Criteria:

* Military personnel ≥17 years of age.
* Completion of the DoD Smallpox Screening Form 600 (2-part format).

Exclusion Criteria:

* None

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This study involves a review of DoD Smallpox Screening Form 600 (2 part format) that had been redacted of all personal information by the DoD. No individuals were involved in this study."
Sampling Method: Non-Probability Sample
Enrollment: 5001 (Actual)
Dates: Start 2009-09; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
The percent of SF600 forms that did not clearly support the subsequent decision to vaccinate. | 1 year post-screening
  ACAM2000® Screening Accuracy Review Committee (SARC) consensus that SF600 form did not support the decision to vaccinate divided by all subjects in the Evaluable Population.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Emergent BioSolutions
Locations (1):
- Alexandria, Virginia, United States